CLINICAL TRIAL: NCT04715464
Title: Active Surveillance Cultures for Multidrug Resistant Gram-Negative Organisms at an Acute Care Hospital
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 023.PHA.2015.C
Record Dates: First submitted 2019-04-03; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2019-04

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: review of surveillance cultures within the past year — ASC results are reported as positive or negative based on the culture source. Antimicrobial susceptibility testing is performed but not reported; however, physicians may obtain susceptibility information for MDR GNB only if clinically indicated through the microbiology department.
  1. Nasal swab for MRSA
  2. Respiratory specimens
  i. Sputum for MRSA, VRE, and Multi Drug Resistant gram-negative Bacteria (MDR GNB) (if not intubated but with productive cough) ii. Endotracheal aspirate for MRSA, VRE, and MDR GNB (if intubated) c. Drainage from any wounds for MRSA, VRE, and MDR GNB d. Rectal/ perianal swab for VRE, and MDR GNB e. Urine for MRSA, VRE, and MDR GNB (from patients catheterized prior to admission only)

SUMMARY:
Active Surveillance Culture programs (ASC) have been initiated in health-care systems in recent years as a mechanism for tracking multi-drug resistant organisms (MDRO), with a goal to reduce the transfer of those organisms to other patients. Consequently, the Center for Disease Prevention and Control (CDC) charged infection control personnel to develop institutional guidelines for the prevention of transmission of multidrug-resistant organisms, within health care settings. The CDC guidelines include performance of active surveillance cultures for patients after admission to health care facilities or to high-risk-patient care units, to detect colonization with target multidrug-resistant organisms. The most commonly tracked antimicrobial resistance organisms in hospital surveillance programs are methicillin resistant Staphylococcus aureus (MRSA), vancomycin resistant enterococcus (VRE), Clostridium difficile, extended-spectrum beta-lactamase (ESBL) producing gram-negative bacilli (e.g. Escherichia coli, Klebsiella pneumoniae), and carbapenem resistant Enterobacteriaceae (CRE). Patients who are colonized with these potential pathogens are placed under contact precautions to prevent transmission to other patients. While clinical outcomes studies exist for MDR gram-positive organisms [particularly methicillin resistant Staphylococcus aureus (MRSA)] ASC, data is limited for MDR gram-negative organisms. The study is retrospective cohort study to evaluate if isolation of an MDR gram-negative pathogen on ASC predicts subsequent infection with the same pathogen.

Patients >18 years of age, admitted to MHS with ASC for MDR gram-negative pathogens, will be included if criteria met. Outcomes of interest will be evaluated with appropriate statistical tests, and multivariate analyses will be used to control for predictors of interest. All analysis will be considered significant at an alpha of <0.05. The investigators anticipate that increased screening with isolation will result in decreased subsequent MDRO gram-negative infection. Furthermore, the investigators hope that this will also result in improved patient's outcomes, mortality, and decreased cost, including excessive use of anti-infectives and its unintended consequences such as microbial resistance.

DETAILED DESCRIPTION:
This is a retrospective cross-sectional study of patients with ASC at MHS. Patients >18 years of age, admitted to MHS during the study specified period, will be included if there is documented ASC. Patients will be identified through the clinical microbiology laboratory records. Figure 1 is a flow diagram of ASC stratification.

Study populations All patients with documented laboratory surveillance culture from January 1, 2006 to December 31, 2012 will be included. Eligible cultures (see definitions below) will be identified based on positive surveillance cultures from MHS. Patients identified with select criteria per objective will be further analyzed in subsequent phases to complete all outcomes of interest. Patients will be excluded if they are ≤18 years, expired before initial surveillance culture is positive, were not admitted, or were transferred to another institution. Patients will be excluded if they underwent amputation or surgical revision for wound infections. Patients with polymicrobial MDR gram-negative pathogen on ASC will be included; however, the main focus of this study is the subset of patients with monomicrobial ASC. Lastly, only the index culture will be considered, for patients with multiple wounds ASC.

Data Collection Initial phase will focus on review of surveillance cultures within the past year (calendar year 2012) to determine objective number one. Prior years are included to evaluate earlier documentation of colonization and whether number of patients/cultures per year has significant variation. Subsequent phases will collect specific data identified as significant or varied based on previous analysis. Data will be collected via extraction and chart review from MHS's electronic medical record (EMR) on identified patients.

Patient demographics (weight, sex, race, age, allergy), co-morbid conditions (diabetes, immunosuppressed, HIV/AIDS, organ transplant, malignancy, chronic lung disease, chronic kidney disease, liver disease, surgery in past 30 days), location in the hospital, type of residence (i.e., home, long-term care facility, etc), source of infection, treatment data (antibiotics administered and duration), length of stay in survivors, hospital cost, antibiotic cost, severity of illness by mean Simplified Acute Physiologic Score (SAPS) II score (based on clinical data present during the 24 hours preceding the index blood culture), hospital mortality, and DRG. Previous hospitalizations, antimicrobial usage and surveillance culture results will be recorded.

Surveillance cultures from nares, rectum, endotracheal aspirates, urine, and wound swab will be included. Microbiology data (organism, culture source, and number of classes of antibiotics with resistance) will be documented. Patients with positive ASC for MDR gram-negative pathogens will be evaluated for antimicrobial use for 1) ASC only and 2) Subsequent positive cultures due to suspected or proven active infection. Cost for each of the following classifications will be determined and compared: microbiological cultures including antimicrobial susceptibility test, length of stay, cost of antimicrobial and associated diagnosis related groups (DRG) per infection type.

ELIGIBILITY:
Inclusion Criteria:

* Any inpatient, except patients admitted through Labor & Delivery departments, meeting the following criteria will be cultured
* Patient has one of the following risk factors for MDROs:
* Hospitalization for 2 consecutive nights or more in the preceding 30 days
* Residence in a nursing home or extended/long term care facility
* Presence of decubitus ulcer or a draining wound
* Admission assessment in the Emergency Department and on nursing units includes questions regarding past history of Multi Drug Resistant (MDR) infection or colonization.

Exclusion Criteria

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any inpatient, except patients admitted through Labor & Delivery departments at Methodist Charlton Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 2878 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Positive ASC with an MDR gram-negative pathogen is a predictor of subsequent active infection | January 1, 2006 to December 31, 2012
  development of infection during hospital stay (days)

SECONDARY OUTCOMES:
The extent of antimicrobial treatment secondary to positive ASC | January 1, 2006 to December 31, 2012
  The relationship between antimicrobial usage and increased resistance will decide the cost of treatment (dollars)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Akins, PharmD, Principal Investigator — Methodist Health System